CLINICAL TRIAL: NCT06208865
Title: Association of Fatty Infiltration in Paraspinal Muscles With the Analgesic Effect of Lumbar Erector Spina Plane Block
Brief Title: Fatty Infiltration in Paraspinal Muscles and Lumbar Erector Spina Plane Block
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Medical doctor, Diskapi Teaching and Research Hospital
Other Study IDs: Lumbar ESPB
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
Keywords: plane block; low back pain; lumbar radiculopathy; fatty infiltration; erector spinae muscles
MeSH Terms: conditions — Low Back Pain; Radiculopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lumbar erector spinae plane block — All procedures were performed under ultrasound (US) guidance. The patient was monitored in the operating room and placed in the prone position under a sterile drape. A 2-6 MHz convex US probe was used during the procedure. The transverse processes of the lumbar vertebrae were visualized and then a 22 gauge spinal needle was advanced to the transverse process of the L3 vertebra. After contacting the transverse process, a total of 15 mL of drug consisting of 2 mL of methylprednisolone and 6 mL of 0.025% bupivacaine was injected into this area, and the spread of the drug in the craniocaudal area was visualized. The patients were followed up for possible complications after the procedure.

SUMMARY:
This study aimed to investigate the relationship between fatty infiltration in the lumbar paraspinal (multifidus and erector spinae) muscles, clinical characteristics, and treatment response after lumbar erector spinae plane block (ESPB) in patients with low back pain due to lumbar radiculopathy. A responder was defined as a patient with a numerical rating scale (NRS) decrease of ≥ 50% from baseline to one month after the procedure. The presence of fat infiltration in the lumbar paraspinal muscles was assessed, along with patient demographic and clinical characteristics.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common health problem that causes global disability. Lumbosacral radiculopathy (LR) is the most common cause of low back pain. Disc herniation is the most common cause of LR, in addition to spinal stenosis, foraminal stenosis, facet joint hypertrophy, and degenerative disease (1). Treatment options for lumbar disc herniation include conservative treatment, interventional pain management, and surgery. Lumbar erector spinae plane block (ESPB) is an interventional procedure for chronic axial and radicular low back pain which that is unresponsive to conservative treatment.

Lumbar paraspinal muscles play an important role in maintaining lumbar spine stability. Increased fat infiltration in the paraspinal muscles has been associated with high-intensity low back pain and poor functional status, and fat infiltration in the paraspinal muscles can be detected by lumbar magnetic resonance imaging. In this study, fatty infiltration in the bilateral lumbar multifidus muscles was evaluated at the L3 level using Goutallier classification.

The primary aim of this study was to investigate the potential relationship between the treatment outcome of lumbar ESPB and the degree of fatty infiltration in the paraspinal muscles in patients with chronic axial and/or radicular low back pain unresponsive to conservative treatments. The secondary aim was to identify other factors that may be associated with a successful response to lumbar ESPB and fatty infiltration of the paraspinal muscles.

ELIGIBILITY:
Inclusion Criteria:

* lumbar radicular pain
* no response to conservative treatment for > 3 months
* MRI within 1 year prior to injection.

Exclusion Criteria:

* inadequate medical records with missing numerical rating scale (NRS) scores and MRI images
* patients lost to follow-up within one month after lumbar ESPB
* patients with a history of surgery for lumbar disc herniation
* patients with severe spinal and/or foraminal stenosis
* patients with extruded, sequestrated, or migrating hernias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male and female patients who underwent lumbar erector spinae plane block for low back pain due to lumbar radiculopathy
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
VAS | Change from Baseline NRS at 3 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, MD, Principal Investigator — Diskapi Teaching and Research Hospital; Ezgi Can, MD, Study Director — Diskapi Teaching and Research Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided